CLINICAL TRIAL: NCT06984003
Title: Efficacy of Pulsed Electromagnetic Field Versus Active Stretching Exercises on Primary Dysmenorrhea
Brief Title: Pulsed Electromagnetic Field Versus Active Stretching Exercises on Primary Dysmenorrhoea Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rabab Ali Mohamed, Assistant Professor of Physical Therapy, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (P.T. REC/012/005704)
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Pulsed Electromagnetic Field; Active Stretching Exercises
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulsed electromagnetic (Experimental): The magnetotherapy device (level s.r.l. SEDE LEGALE, Catania, Italia) consists of the control panel, motorized bed, and two solenoids (52 cm in diameter for the stand and 80 cm in diameter for the bed). The control panel is connected to electrical mains, supplying 230 V AC 50 Hz. graphic display, multifunction control with encoder selection through a MENU SUBMENU, making the machine easy to use. Pillows and cushions were used to support body parts in a comfortable, relaxed position, and sheets were used to cover the patients during treatment sessions. Participants randomly assigned into Group A (n = 15) received PEMF applied to the pelvic region 3 days per week for 8 weeks, twenty minutes per day. The used parameters of PEMF were 50 Hz in frequency and 60 G in intensity applied in the comfortable supine lying position with small pillows under the participants' body curves.
  Interventions: Other: stretching exercises

INTERVENTIONS:
Other: stretching exercises — a brief explanation, by a trained physical therapist, of stretching exercise program and of how to practice these active stretching exercises as a home program 3 times per week for 4 weeks.

SUMMARY:
Primary dysmenorrhea (PD) refers to painful cramps before and/or during menstruation. There is a need for emphasis on alternative methods of conservative treatment, so as to reduce the dependence on drugs for alleviating the symptoms., so the aim of this study was to investigate the effect of pulsed electromagnetic field versus active Stretching exercises on primary dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea is a menstrual disorder characterized by suprapubic cramping of uterine origin and pain occurring a few hours before or after the onset of menstruation. Primary dysmenorrhea begins when young girls experience the first menstrual adulatory cycles, and its prevalence increases during adolescence (15-17 years) and reaches its highest at 20-24 years and decreases progressively thereafter. Primary dysmenorrhea is characterized by abdominal pain, beginning a few hours before and continuing up to 12-72 hours, and is like the delivery of pains along with cramps in the lower abdomen radiating toward the inner side of the thighs. Half of such cases experience systemic symptoms, such as nausea, vomiting, diarrhea, fatigue, irritability, and dizziness.

Primary dysmenorrhea occurs in up to 50% of menstruating females and causes significant disruption in quality of life.4 Menstrual cramps are associated with nausea in 55% and with vomiting in 24%.5 The severity of symptoms positively correlates with the onset of ovulatory cycles and with increased duration and amount of menstrual flow.6 A physiological reason for dysmenorrhea is the production of uterine prostaglandins. During endometrial sloughing, endometrial cells release prostaglandins as menstruation begins. Prostaglandins stimulate myometrial contractions and ischemia.7 During the recent 20-30 years, regular exercise and physical activities have been introduced as effective methods for prevention and treatment of dysmenorrhea.8Exercising affects the levels of steroid hormones in the blood circulation of women in reproductive ages.9 Moreover, the elevation of the endorphin hormone leads to an increase in pain threshold.10 Pulsed electromagnetic field (PEMF) is an efficient modality used in physical therapy field for treatment of many pathological cases; PEMF has strong analgesic effect, anti-inflammatory effect, and a vasodilatation effect, as well as decreasing edema.11 PEMF has electric energy and generates series of magnetic pulses through the tissues, and each magnetic pulse induces a tiny electrical signal that stimulates cellular repair, suppresses inflammatory responses, alleviates pain, and increases range of motion.12 PEMF are effective in relieving pain of primary dysmenorrhea by decreasing prostaglandin levels in the blood, resulting in fewer vigorous uterine contractions and less discomfort.

A range of treatment options have been examined in the literature, including heat application, pelvic floor and aerobic exercises, low-level laser therapy, and pulsed electromagnetic field, with several producing effective outcomes. These interventions were assumed to prevent or minimize menstrual pain by increasing pelvic circulation, decreasing uterine contractions, and activating the release of endorphins and serotonin, but there is still no evidence for the best type of modality chosen.

Additional researches are needed to clarify difference between effect of Pulsed electromagnetic field (PEMF) and active stretching on pain intensity level and menstrual symptoms in females with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Young female students suffering from primary dysmenorrhea
* regular menstrual cycle diagnosed by gynecologist
* BMI ranging from 18.5 to 25 kg/ m 2.
* Pain intensity is 4 or above in VAS.
* Their ages ranged from 18- 24 years old-

Exclusion Criteria:

* Girls with irregular or infrequent menstrual cycles, using pharmacological or non-pharmacological methods for pain relief during the study
* suffering from pelvic pathology

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
pain intensity assessment in primary dysmenorrhea | 4 weeks
  by using a visual analogue scale (VAS) was performed before and after the treatment. VAS is a self-reported 10-cm straight line, which represents the pain intensity, with the two opposite ends representing no pain and worst pain. Based on the VAS scale, those subjects with pain intensity of 4 to 7 were classified as the moderate group. The subjects with a pain score between 7 and 10 were considered to have a severe form of dysmenorrhea. The subjects with pain intensity less 4 were excluded from the research design. Each participant was asked to place a mark along the line to denote the level of pain

CONTACTS AND LOCATIONS:
Overall Officials: Rabab Ali Mohamed, PHD, Principal Investigator — Cairo University Faculty of Physical Therapy; Rabab A Mohamed, PHD, Principal Investigator — Basic Science Department, Faculty of Physical Therapy, Cairo University, Egypt. 2Department of Physical Therapy, College of Applied Medical Sciences, Qassim University, Buraidah 51452, Saudi Arabia.
Locations (1):
- Faculty of Physical Therapy, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No